CLINICAL TRIAL: NCT03610334
Title: A Double-blind, Randomized, Placebo-controlled, Combined Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability and Pharmacokinetic Profile of IFB-088, in Healthy Volunteers
Brief Title: A Combined SAD and MAD Study to Investigate the Safety, Tolerability and Pharmacokinetic Profile of IFB-088
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InFlectis BioScience (Industry)
Collaborators: Qualissima (Other); Assistance Publique Hopitaux De Marseille (Other); Stragen France (Industry); Eurofins Optimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: P188; 2018-000443-29 (EudraCT Number)
Record Dates: First submitted 2018-06-20; First posted 2018-08-01 (Actual); Results first posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-11

CONDITIONS: Healthy Volunteers
Keywords: First-In-Human
MeSH Terms: interventions — calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Intervention Model Description: double-blind, randomized, placebo-controlled, combined single and multiple ascending dose of IFB-088 by successive cohorts study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Capsules used for verum or placebo (Size 5 white opaque HPMC capsule) are identical and equally-weighted
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- SAD IFB-088 2.5mg (Experimental): Cohort 1: A single daily dose of 2.5mg IFB-088 in oral capsule, is administered with 250 ml of water at room temperature, in the morning around 8:00am, in one intake
  Interventions: Drug: IFB-088 (2.5-60.0mg) oral capsule
- SAD Placebo 2.5mg (Placebo Comparator): Cohort 1: A single daily dose of 2.5mg placebo in oral capsule, is administered with 250 ml of water at room temperature, in the morning around 8:00am, in one intake
  Interventions: Drug: Placebo (2.5-60.mg) oral capsule
- SAD IFB-088 5.0mg (Experimental): Cohort 2: A single daily dose of 5.0mg IFB-088 in oral capsule, divided in two doses of 2.5mg are administered with 250 ml of water at room temperature, seperated by an interval of 12h, in the morning around 8:00am, and in the evening around 8:00pm
  Interventions: Drug: IFB-088 (2.5-60.0mg) oral capsule
- SAD Placebo 5.0mg (Placebo Comparator): Cohort 2: A single daily dose of 5.0mg placebo in oral capsule, divided in two doses of 2.5mg are administered with 250 ml of water at room temperature, seperated by an interval of 12h, in the morning around 8:00am, and in the evening around 8:00pm
  Interventions: Drug: Placebo (2.5-60.mg) oral capsule
- SAD IFB-088 10.0mg (Experimental): Cohort 3: A single daily dose of 10.0mg IFB-088 in oral capsule, divided in two doses of 5.0mg are administered with 250 ml of water at room temperature, seperated by an interval of 12h, in the morning around 8:00am, and in the evening around 8:00pm
  Interventions: Drug: IFB-088 (2.5-60.0mg) oral capsule
- SAD Placebo 10.0mg (Placebo Comparator): Cohort 3: A single daily dose of 10.0mg Placebo in oral capsule, divided in two doses of 5.0mg are administered with 250 ml of water at room temperature, seperated by an interval of 12h, in the morning around 8:00am, and in the evening around 8:00pm
  Interventions: Drug: Placebo (2.5-60.mg) oral capsule
- SAD IFB-088 20.0mg (Experimental): Cohort 4: A single daily dose of 20.0mg IFB-088 in oral capsule, divided in two doses of 10.0mg are administered with 250 ml of water at room temperature, seperated by an interval of 12h, in the morning around 8:00am, and in the evening around 8:00pm
  Interventions: Drug: IFB-088 (2.5-60.0mg) oral capsule
- SAD Placebo 20.0mg (Placebo Comparator): Cohort 4: A single daily dose of 20.0mg Placebo in oral capsule, divided in two doses of 10.0mg are administered with 250 ml of water at room temperature, seperated by an interval of 12h, in the morning around 8:00am, and in the evening around 8:00pm
  Interventions: Drug: Placebo (2.5-60.mg) oral capsule
- SAD IFB-088 40.0mg (Experimental): Cohort 5: A single daily dose of 40.0mg IFB-088 in oral capsule, divided in two doses of 20.0mg are administered with 250 ml of water at room temperature, seperated by an interval of 12h, in the morning around 8:00am, and in the evening around 8:00pm
  Interventions: Drug: IFB-088 (2.5-60.0mg) oral capsule
- SAD Placebo 40.0mg (Placebo Comparator): Cohort 5: A single daily dose of 40.0mg Placebo in oral capsule, divided in two doses of 20.0mg are administered with 250 ml of water at room temperature, seperated by an interval of 12h, in the morning around 8:00am, and in the evening around 8:00pm
  Interventions: Drug: Placebo (2.5-60.mg) oral capsule
- SAD IFB-088 60.0mg (Experimental): Cohort 6: A single daily dose of 60.0mg IFB-088 in oral capsule, divided in two doses of 30.0mg are administered with 250 ml of water at room temperature, seperated by an interval of 12h, in the morning around 8:00am, and in the evening around 8:00pm
  Interventions: Drug: IFB-088 (2.5-60.0mg) oral capsule
- SAD Placebo 60.0mg (Experimental): Cohort 6: A single daily dose of 60.0mg Placebo in oral capsule, divided in two doses of 30.0mg are administered with 250 ml of water at room temperature, seperated by an interval of 12h, in the morning around 8:00am, and in the evening around 8:00pm
  Interventions: Drug: Placebo (2.5-60.mg) oral capsule
- MAD IFB-088 15 mg (Experimental): Cohort 7: subject taking 15.0mg of IFB-088 in oral capsule divided into 2 doses of 7.5mg administered with 250ml of water at room temperature, seperated by an interval of 12h, in the morning around 8:00am, an in the evening around 8:00pm, for 14 days.
  Interventions: Drug: IFB-088 (15.0-50.0mg) oral capsule
- MAD Placebo 15 mg (Placebo Comparator): Cohort 7: subject taking 15.0mg of placebo in oral capsule divided into 2 doses of 7.5mg administered with 250ml of water at room temperature, seperated by an interval of 12h, in the morning around 8:00am, an in the evening around 8:00pm, for 14 days.
  Interventions: Drug: Placebo oral (15.0-50.0mg) capsule
- MAD IFB-088 30 mg (Experimental): Cohort 8: subject taking 30.0mg of IFB-088 in oral capsule divided into 2 doses of 15.0mg administered with 250ml of water at room temperature, seperated by an interval of 12h, in the morning around 8:00am, an in the evening around 8:00pm, for 14 days.
  Interventions: Drug: IFB-088 (15.0-50.0mg) oral capsule
- MAD Placebo 30 mg (Placebo Comparator): Cohort 8: subject taking 30.0mg of Placebo in oral capsule divided into 2 doses of 15.0mg administered with 250ml of water at room temperature, seperated by an interval of 12h, in the morning around 8:00am, an in the evening around 8:00pm, for 14 days.
  Interventions: Drug: Placebo oral (15.0-50.0mg) capsule
- MAD IFB-088 50 mg (Experimental): Cohort 9: subject taking 50.0mg of IFB-088 in oral capsule divided into 2 doses of 25.0mg administered with 250ml of water at room temperature, seperated by an interval of 12h, in the morning around 8:00am, an in the evening around 8:00pm, for 14 days.
  Interventions: Drug: IFB-088 (15.0-50.0mg) oral capsule
- MAD Placebo 50 mg (Placebo Comparator): Cohort 9: subject taking 50.0mg of Placebo in oral capsule divided into 2 doses of 25.0mg administered with 250ml of water at room temperature, seperated by an interval of 12h, in the morning around 8:00am, an in the evening around 8:00pm, for 14 days.
  Interventions: Drug: Placebo oral (15.0-50.0mg) capsule

INTERVENTIONS:
Drug: IFB-088 (2.5-60.0mg) oral capsule — SAD phase: IFB-088 will be administered during 1 day, in one (2.5mg) or 2 (5.0-60.0mg) intakes separated by an interval of 12 hours
  Other Names: verum
  Arms: SAD IFB-088 10.0mg; SAD IFB-088 2.5mg; SAD IFB-088 20.0mg; SAD IFB-088 40.0mg; SAD IFB-088 5.0mg; SAD IFB-088 60.0mg
Drug: Placebo (2.5-60.mg) oral capsule — SAD phase: placebo (microcrystalline cellulosis) will be administered during 1 day, in one (2.5mg) or 2 (5.0-60.0mg) intakes separated by an interval of 12 hours
  Other Names: placebo
  Arms: SAD Placebo 10.0mg; SAD Placebo 2.5mg; SAD Placebo 20.0mg; SAD Placebo 40.0mg; SAD Placebo 5.0mg; SAD Placebo 60.0mg
Drug: IFB-088 (15.0-50.0mg) oral capsule — MAD phase: multiple doses of IFB-088 (15.0-50.0mg) will be administered daily during 14 days, in two intakes, separated by an interval of 12 hours.
  Other Names: verum
  Arms: MAD IFB-088 15 mg; MAD IFB-088 30 mg; MAD IFB-088 50 mg
Drug: Placebo oral (15.0-50.0mg) capsule — MAD phase: multiple doses of placebo (microcrystalline cellulosis, 15.0-50.0mg) will be administered daily during 14 days, in two intakes, separated by an interval of 12 hours.
  Other Names: placebo
  Arms: MAD Placebo 15 mg; MAD Placebo 30 mg; MAD Placebo 50 mg

SUMMARY:
This is the first study of single and multiple doses of IFB-088 in human subjects. The current study is designed to assess in the first part, the safety, tolerability, plasma and urine pharmacokinetics (PK) of single oral doses of IFB-088 in healthy subjects (Single Ascending Doses - SAD) and in a second part safety, tolerability, plasma and urine pharmacokinetics (PK) of multiple oral doses of IFB-088 in healthy subjects (Multiple Ascending Doses - MAD)

DETAILED DESCRIPTION:
Randomized, double blind, placebo controlled study of single ascending doses (SAD) and multiple ascending doses (MAD).

The SAD part consists of 6 cohorts of 8 healthy young male subjects, each receiving a single oral dose of IFB-088 or placebo (6 verum and 2 placebo). In each cohort, 2 subjects (1 verum and 1 placebo) will be dosed first. If the safety and tolerability results are acceptable, the 6 remaining subjects will be dosed by 2 successive groups of 3 subjects, with an adequate period between the 2 groups to detect the occurrence of any reaction or adverse events, namely at least 48H for the first cohort and at least 36H for the following cohorts. Indeed, in the first cohort (2.5 mg IFB-088 base), dosing will be in the morning only. From the second cohort, the planned daily dose will be divided into 2 doses separated by an interval of 12 hours (1 dose in the morning fasting and 1 dose in the evening 2 hours before dinner).

The MAD part consists of 3 cohorts of 8 healthy young male subjects, each receiving an oral dose divided into two doses of IFB-088 or placebo (6 verum and 2 placebo) for 14 days. In each cohort, the 2 first subjects will be dosed on Day 1 (one on active treatment and one on placebo). The 6 remaining subjects will be dosed by 2 successive groups of maximum 3 subjects with an adequate period between the groups to observe for any reaction and adverse events. This period will be of at least 36H, corresponding to at least 5-fold the half-life of the drug (based on results obtained during the SAD part) when steady state will be achieved. In each MAD cohort, the total daily dose will be divided into 2 doses separated by an interval of 12 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male 18 to 40 years of age inclusive, Caucasian.
2. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests, vital signs and ECG.
3. AST, ALT, alkaline phosphatase and bilirubin < or = 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
4. ECG (12 leads) normal (120<PR<200ms; QRS<120ms; QTcF<450ms) and/or without clinically relevant impairments as judged by investigator.
5. Non-smoker, or user of not more than tobacco- or nicotine-containing products ≤ 5 cigarettes a day.
6. Negative screen for alcohol and drugs of abuse at screening and admission.
7. No history of psychiatric disorders assessed by a clinical psychological evaluation and the Mini International Neuropsychiatric Interview (MINI).
8. Body mass index (BMI) between 19 and 27 kg/m² inclusive.
9. Subject with female partners of child bearing potential must agree to use one of the contraception methods listed in Section 6.6.1 (Contraception requirements). This criterion must be followed from the time of the first dose of study medication until the follow up visit (for female partners) and with an additional period of 90 days (for subjects themselves).
10. Willing and able to understand and sign an approved Informed Consent Form.
11. Able to understand the protocol and to come to the visits.
12. Who is, in the judgement of the investigator likely to be compliant during the study.
13. Subject registered in the VRB file (volontaires se prêtant à des recherches impliquant la personne humaine).
14. Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research.

Exclusion Criteria:

1. 1. History of asthma, anaphylaxis or anaphylactoid reactions, severe allergic responses.
2. History of relevant atopy or drug hypersensitivity.
3. Known allergy to any component of IFB-088 oral capsule or its placebo (HPMC or cellulose microcrystalline).
4. History of major medical, psychiatric illness or surgery which, in the judgment of the investigator, puts them 'at risk' or is likely to modify their handling of the study drug.
5. Acute or chronic systemic disease or disorder (respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine).
6. Impaired renal function defined by a creatinine clearance < 90 mL/min calculated using the Cockcroft-Gault equation (according the FDA Guidance for Industry: Pharmacokinetics in patients with Impaired Renal Function, March 2010).
7. History of nephritic colic and/or renal calculi.
8. History of drug abuse and/or regular use of tobacco- or nicotine-containing products > 5/day within three months of the study.
9. History of alcohol consumption exceeding, (on average 21 drinks/week for men) within 6 months of the first dose of study medication.
10. Drinking excessive amounts of tea, coffee, chocolate and/or beverage containing caffeine (> 4 cups / day).
11. Vital signs with a clinically significant abnormality at screening.
12. ECG with a clinically significant abnormality at screening.
13. Laboratory test values outside the clinically acceptable 'normal range' for healthy volunteers at screening.
14. Positive HIV, Hepatitis B or Hepatitis C at screening.
15. Positive urine drug test or positive breath alcohol test at screening or at admission to the clinical unit.
16. Any medication (including St John's Wort) within 14 days before administration, or within 5 times the elimination half-life of that drug, whichever is the longest (except paracetamol).
17. Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to screening.
18. Unable to refrain from consumption of grapefruit or grapefruit juice within 7 days prior to the first dose of study medication.
19. Unwillingness to abstain from sexual intercourse with pregnant or lactating women or to use a condom and spermicide and another form of contraception (e.g., IUD, birth control pills taken by female partner, diaphragm with spermicide) if engaging in sexual intercourse with a woman who could become pregnant until discharge from the study and during 90 additional days.
20. Subjects unlikely to co-operate in the study, and/or poor compliance anticipated by the investigator.
21. Subject being in the exclusion period of a previous trial.
22. Subject having exceeded the earnings for the last 12 months, including the indemnities for the present study.
23. Subject who could not be contacted in case of emergency.
24. Subject refusing to give written informed consent.
25. Subject who has received blood or plasma derivatives in the year preceding the study.
26. Subject who has given blood within the past 3 months or has planned to give blood or sperm within the 90 days following the study.
27. Subject who has forfeited their freedom by administrative or legal award, or who is under guardianship or under limited judicial protection.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Audebert, MD, Principal Investigator — APHM - Centre de Pharmacolgie Clinique et d'Evaluations Thérapeutiques
Locations (2):
- France (2):
  - Eurofins|Optimed, Gières
  - Centre d'Investigation Clinique - Centre de Pharmacologie Clinique et d'Evaluations Thérapeutiques (CIC-CPCET), Marseille

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of InFlectis BioScience — http://www.inflectisbioscience.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- SAD IFB-088 2.5 mg: A single daily dose of IFB-088 2.5 mg is administered to 6 healthy volunteers
- SAD Placebo 2.5mg: A single daily dose of placebo (microcristalline cellusose) 2.5 mg is administered to 2 healthy volunteers
- SAD IFB-088 5.0mg: Administration of the drug to this group of new healthy volunteers is conditionned to the safety obtained in the previous period.
  A single daily dose of IFB-088 5.0 mg is administered to 6 healthy volunteers, in two intakes of 2.5mg, separated by 12h.
- SAD Placebo 5.0mg: Administration of the placebo to this group of new healthy volunteers is conditionned to the safety obtained in the previous period.
  A single daily dose of placebo (microcrystalline cellulose) 5.0 mg is administered to 2 healthy volunteers, in two intakes of 2.5mg, separated by 12h.
- SAD IFB-088 10.0mg: Administration of the drug to this group of new healthy volunteers is conditionned to the safety obtained in the previous period.
  A single daily dose of IFB-088 10.0 mg is administered to 6 healthy volunteers, in two intakes of 5.0mg, separated by 12h.
- SAD Placebo 10.0mg: Administration of the placebo to this group of new healthy volunteers is conditionned to the safety obtained in the previous period.
  A single daily dose of placebo (microcrystalline cellusose) 10.0 mg is administered to 2 healthy volunteers, in two intakes of 5.0mg, separated by 12h.
- SAD IFB-088 20.0mg: Administration of the drug to this group of new healthy volunteers is conditionned to the safety obtained in the previous period.
  A single daily dose of IFB-088 20.0 mg is administered to 6 healthy volunteers, in two intakes of 10.0mg, separated by 12h.
- SAD Placebo 20.0mg: Administration of the placebo to this group of new healthy volunteers is conditionned to the safety obtained in the previous period.
  A single daily dose of placebo (microcrystalline cellusose) 20.0 mg is administered to 2 healthy volunteers, in two intakes of 10.0mg, separated by 12h.
- SAD IFB-088 40.0mg: Administration of the drug to this group of new healthy volunteers is conditionned to the safety obtained in the previous period.
  A single daily dose of IFB-088 40.0 mg is administered to 6 healthy volunteers, in two intakes of 20.mg, separated by 12h.
- SAD Placebo 40.0mg: Administration of the placebo to this group of new healthy volunteers is conditionned to the safety obtained in the previous period.
  A single daily dose of placebo (microcrystalline cellusose) 40.0 mg is administered to 2 healthy volunteers, in two intakes of 20.0mg, separated by 12h.
- SAD IFB-088 60.0mg: Administration of the drug to this group of new healthy volunteers is conditionned to the safety obtained in the previous period.
  A single daily dose of IFB-088 60.0 mg is administered to 6 healthy volunteers, in two intakes of 30.0mg, separated by 12h.
- SAD Placebo 60.0mg: Administration of the placebo to this group of new healthy volunteers is conditionned to the safety obtained in the previous period.
  A single daily dose of placebo (microcrystalline cellusose) 60.0 mg is administered to 2 healthy volunteers, in two intakes of 30.0mg, separated by 12h.
- MAD IFB-088 15.0mg: Administration of the drug to this group of new healthy volunteers is conditionned to the safety obtained in the Single Ascending Dose Study.
  A single dose of IFB-088 15.0 mg is administered to 6 healthy volunteers, during 14 days
- MAD Placebo 15.0mg: Administration of the placebo to this group of new healthy volunteers is conditionned to the safety obtained in the Single Ascending Dose Study.
  A single dose of placebo (microcrystalline cellulose) 15.0 mg is administered to 2 healthy volunteers, during 14 days
- MAD IFB-088 30.0mg: Administration of the drug to this group of new healthy volunteers is conditionned to the safety obtained in the previous period.
  A dose of IFB-088 30.0 mg is administered in two intakes of 15.0mg, administered at 12hours of interval, to 6 healthy volunteers, during 14 days.
- MAD Placebo 30.0mg: Administration of the placebo to this group of new healthy volunteers is conditionned to the safety obtained in the previous period.
  A dose of placebo (microcrystalline cellulose) 30.0 mg is administered in two intakes of 15.0mg, administered at 12hours of interval, to 2 healthy volunteers, during 14 days.
- MAD IFB-088 50.0mg: Administration of the drug to this group of new healthy volunteers is conditionned to the safety obtained in the previous period.
  A dose of IFB-088 50.0 mg is administered in two intakes of 25.0mg, administered at 12hours of interval, to 6 healthy volunteers, during 14 days.
- MAD Placebo 50.0mg: Administration of the placebo to this group of new healthy volunteers is conditionned to the safety obtained in the previous period.
  A dose of placebo (microcrystalline cellulose) 50.0 mg is administered in two intakes of 25.0mg, administered at 12hours of interval, to 2 healthy volunteers, during 14 days.
Period: Period 1: 2.5mg (1 Day)
Arm/Group | SAD IFB-088 2.5 mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Started | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2: 5.0mg (1 Day)
Arm/Group | SAD IFB-088 2.5 mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Started | 6 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3: 10.0mg (1 Day)
Arm/Group | SAD IFB-088 2.5 mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Started | 6 | 2 | 6 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 2 | 6 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4: 20.0mg (1 Day)
Arm/Group | SAD IFB-088 2.5 mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Started | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5: 40.0mg (1 Day)
Arm/Group | SAD IFB-088 2.5 mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Started | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 6: 60.0mg (1 Day)
Arm/Group | SAD IFB-088 2.5 mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Started | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 7: 15.0mg (Day 1 to 14)
Arm/Group | SAD IFB-088 2.5 mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Started | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 0 | 0 | 0 | 0
Completed | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 8: 30.0mg (Day 1 to 14)
Arm/Group | SAD IFB-088 2.5 mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Started | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 0 | 0
Completed | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 9: 50.0mg (Day 1 to 14)
Arm/Group | SAD IFB-088 2.5 mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Started | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Completed | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: the trial is divided into 2 phases (SAD and MAD). SAD included a total of 6 cohorts (total of 48 volunteers), with 36 (6x6) volunteers receiving the verum at dose ranging from 2.5mg to 60.0mg/day, and 12 (6x2) receiving the equivalent placebo. MAD included a total of 3 cohorts (total of 24 volunteeres), with 18 (3x6) receiving the verum at dose ranging from 15 to 50mg/day, and 6 (3x2) receiving the equivalent placebo for 14 days.
  All patients were healthy French caucasian male above 18 years.
Groups:
- Cohort 1: SAD IFB-088 2.5mg: a single daily dose of 2.5mg IFB-088 in oral capsule, is administered in the morning (8:00am), in one intake
- Cohort 2: SAD IFB-088 5.0mg: a single daily dose of 5.0mg IFB-088 in oral capsule, divided into 2 doses of 2.5mg, is administered, separated by an interval of 12h (in the morning (8:00am), and in the evening (8:00pm)
- Cohort 3: SAD IFB-088 10.0mg: a single daily dose of 10.0mg IFB-088 in oral capsule, divided into 2 doses of 5.0mg, is administered, separated by an interval of 12h (in the morning (8:00am), and in the evening (8:00pm)
- Cohort 4: SAD IFB-088 20.0mg: a single daily dose of 20.0mg IFB-088 in oral capsule, divided into 2 doses of 10.0mg, is administered, separated by an interval of 12h (in the morning (8:00am), and in the evening (8:00pm)
- Cohort 5: SAD IFB-088 40.0mg: a single daily dose of 40.0mg IFB-088 in oral capsule, divided into 2 doses of 20.0mg, is administered, separated by an interval of 12h (in the morning (8:00am), and in the evening (8:00pm)
- Cohort 6: SAD IFB-088 60.0mg: a single daily dose of 60.0mg IFB-088 in oral capsule, divided into 2 doses of 30.0mg, is administered, separated by an interval of 12h (in the morning (8:00am), and in the evening (8:00pm)
- Cohort 7: MAD IFB-088 15.0mg: subject taking 15.0mg of IFB-088 in oral capsule, divided into 2 doses of 7.5mg, separated by an interval of 12 hours, in the morning (8:00am), and in the evening (8:00pm), for 14 days
- Cohort 8: MAD IFB-088 30.0mg: subject taking 30.0mg of IFB-088 in oral capsule, divided into 2 doses of 15.0mg, separated by an interval of 12 hours, in the morning (8:00am), and in the evening (8:00pm), for 14 days
- Cohort 9: MAD IFB-088 50.0mg: subject taking 50.0mg of IFB-088 in oral capsule, divided into 2 doses of 25.0mg, separated by an interval of 12 hours, in the morning (8:00am), and in the evening (8:00pm), for 14 days
- SAD Placebo Group: a single daily dose of placebo in oral capsule, divided into 1 or 2 doses equivalent to verum, is administered, separated by an interval of 12h (in the morning (8:00am), and in the evening (8:00pm)
- MAD Placebo Group: subject taking placebo equivalent to the verum dose in oral capsule, divided into 2 doses , separated by an interval of 12 hours, in the morning (8:00am), and in the evening (8:00pm), for 14 days
- Total: Total of all reporting groups
Arm/Group | Cohort 1: SAD IFB-088 2.5mg | Cohort 2: SAD IFB-088 5.0mg | Cohort 3: SAD IFB-088 10.0mg | Cohort 4: SAD IFB-088 20.0mg | Cohort 5: SAD IFB-088 40.0mg | Cohort 6: SAD IFB-088 60.0mg | Cohort 7: MAD IFB-088 15.0mg | Cohort 8: MAD IFB-088 30.0mg | Cohort 9: MAD IFB-088 50.0mg | SAD Placebo Group | MAD Placebo Group | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 72
Age, Continuous [Mean (Full Range); unit: Year] — Population: 2 parts: SAD: 48 subjects and MAD: 24 subjects
  Year
    subject age | 31.0 [25.0 to 39.0] | 25.5 [23.0 to 31.0] | 27.5 [23.0 to 31.0] | 24.7 [18.0 to 30.0] | 24.5 [19.0 to 30.0] | 25.5 [18.0 to 30.0] | 27.0 [22.0 to 36.0] | 31.7 [21.0 to 40.0] | 31.0 [24.0 to 40.0] | 26.5 [18.0 to 39.0] | 31.7 [26.0 to 40.0] | 26.5 [18 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 72
Region of Enrollment [Number; unit: participants]
  France | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 72

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events Per Group
Description: This safety outcome lists the number of subjects experiencing adverse events (AEs), whether not related, possibly or unlikely related to the study treatment.
  As all the parameters are developped in the pharmacovigilance section, please do refer to that section for further details.
Time Frame: SAD & MAD phases: Screening visit to End of study visit (7 to 14 days after last dosing) + 30 days
Population: 72 Healthy volunteers included in the study, from inclusion visit, up to study disclosure visit, were followed for TEAE. As this this study was a first in human dose escalating study, if TEAE occured in a group, they were analysed by an independant safety commity as not related, unlikely related or possibly related to the study drug, to evaluate safety of the drug and allow to raise the dose in the next group.
Measure: Count of Participants; unit: Participants
Groups:
- SAD IFB-088 2.5mg: healthy volunteers received IFB-088 2.5mg once daily, in the morning.
- SAD Placebo 2.5mg: healthy volunteers received placebo 2.5mg once daily, in the morning.
- SAD IFB-088 5.0mg: healthy volunteers received IFB-088 5.0mg once daily, in two doses of 2.5mg, separated by a 12h interval.
- SAD Placebo 5.0mg: healthy volunteers received placebo 5.0mg once daily, in two doses of 2.5mg, separated by a 12h interval.
- SAD IFB-088 10.0mg: healthy volunteers received IFB-088 10.0mg once daily, in two doses of 5.0mg, separated by a 12h interval.
- SAD Placebo 10.0mg: healthy volunteers received placebo 10.0mg once daily, in two doses of 5.0mg, separated by a 12h interval.
- SAD IFB-088 20.0mg: healthy volunteers received IFB-088 20.0mg once daily, in two doses of 10.0mg, separated by a 12h interval.
- SAD Placebo 20.0mg: healthy volunteers received placebo 20.0mg once daily, in two doses of 10.0mg, separated by a 12h interval.
- SAD IFB-088 40.0mg: healthy volunteers received IFB-088 40.0mg once daily, in two doses of 20.0mg, separated by a 12h interval.
- SAD Placebo 40.0mg: healthy volunteers received placebo 40.0mg once daily, in two doses of 20.0mg, separated by a 12h interval.
- SAD IFB-088 60.0mg: healthy volunteers received IFB-088 60.0mg once daily, in two doses of 30.0mg, separated by a 12h interval.
- SAD Placebo 60.0mg: healthy volunteers received placebo 60.0mg once daily, in two doses of 30.0mg, separated by a 12h interval.
- MAD IFB-088 15.0mg: healthy volunteers received IFB-088 15.0mg once daily, in the morning, during 14 days.
- MAD Placebo 15.0mg: healthy volunteers received placebo 15.0mg once daily, in the morning, during 14 days.
- MAD IFB-088 30.0mg: healthy volunteers received IFB-088 30.0mg daily, in two doses of 15.0mg, separated by a 12h. interval, during 14 days.
- MAD Placebo 30.0mg: healthy volunteers received placebo 30.0mg daily, in two doses of 15.0mg, separated by a 12h. interval, during 14 days.
- MAD IFB-088 50.0mg; MAD Placebo 50.0mg: healthy volunteers received IFB-088 50.0mg daily, in two doses of 25.0mg, separated by a 12h. interval, during 14 days.
Arm/Group | SAD IFB-088 2.5mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Participants | 1 | 0 | 1 | 1 | 2 | 0 | 2 | 0 | 2 | 1 | 3 | 0 | 4 | 1 | 1 | 0 | 4 | 1

2. Secondary Outcome: Number of Participants With Change in Concomitant Medications
Description: modification in Concomitant medication(s) occuring during the study (if applicable)
Time Frame: SAD & MAD phases: Continuous (Screening visit to End of study visit (7 to 14 days after last dosing) + 30 days)
Measure: Count of Participants; unit: Participants
Groups:
- MAD IFB-088 15.0mg: healthy volunteers received IFB-088 15.0mg daily, in the morning, during 14 days.
- MAD Placebo 15.0mg: healthy volunteers received placebo 15.0mg daily, in the morning, during 14 days.
- MAD Placebo 30.0mg: healthy volunteers received IFB-088 30.0mg daily, in two doses of 15.0mg, separated by a 12h. interval, during 14 days.
- MAD Placebo 50.0mg: healthy volunteers received placebo 50.0mg daily, in two doses of 25.0mg, separated by a 12h. interval, during 14 days.
Arm/Group | SAD IFB-088 2.5mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Participants
  add-on: acetaminophen 1000mg 1/day | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  add-on: naproxen 550mg bid | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  add-on: fexofenadine 180mg 1/day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  add-on: desloratadine 5 mg as needed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants without change | 6 | 2 | 6 | 2 | 6 | 2 | 5 | 2 | 5 | 2 | 4 | 2 | 5 | 2 | 6 | 2 | 6 | 2

3. Secondary Outcome: Pharmacokinetic: Maximum Observed Plasma Concentration (Cmax)
Description: Plasma samples are collected:
  SAD phase - cohort 1 (one intake for daily administration): Day 1 at predose, 0.16, 0.33, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 24, 32 hours
  SAD phase - cohort 2 to 6 (two intakes for daily administration): Day 1 at predose, 0.33, 0.66, 1, 2, 3, 4, 5, 12, 12.25, 12.5, 13, 14, 16, 18, 24, 32 hours
  MAD phase (two intakes for daily administration): Day 1 and Day 14 at predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 13, 14, 17, 19 and 21h ; Day 2 (24 hours); Day 7 (predose, 1h and 2 h post dose); Day 15 (24, 30, 36 and 42 hours after Day 14); Day 16 (48, 60 hours after Day 14).
Time Frame: Starting 1 hour prior to dosing on Day 1 and until 72 hours after last dosing (Day 17)
Population: 6 patients per cohort have received the verum and are presented. In all groups but one, patients received the verum twice daily. Cmax has hence been measured twice. In the SAD IFB-088 2.5mg cohort, 0 patient received dose 2 as only 1 dose (dose 1) of 2.5mg was given to the patient therefore Cmax Dose 2 has not been measured.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- MAD IFB-088 15.0mg: Cohort 7: subject taking 15.0mg of IFB-088 in oral capsule divided into 2 doses of 7.5mg administered with 250ml of water at room temperature, seperated by an interval of 12h, in the morning around 8:00am, an in the evening around 8:00pm, for 14 days.
  IFB-088 (15.0-50.0mg) oral capsule: MAD phase: multiple doses of IFB-088 (15.0-50.0mg) will be administered daily during 14 days, in two intakes, separated by an interval of 12 hours.
- MAD IFB-088 30.0mg: Cohort 8: subject taking 30.0mg of IFB-088 in oral capsule divided into 2 doses of 15.0mg administered with 250ml of water at room temperature, seperated by an interval of 12h, in the morning around 8:00am, an in the evening around 8:00pm, for 14 days.
  IFB-088 (15.0-50.0mg) oral capsule: MAD phase: multiple doses of IFB-088 (15.0-50.0mg) will be administered daily during 14 days, in two intakes, separated by an interval of 12 hours.
- MAD IFB-088 50.0mg: Cohort 9: subject taking 50.0mg of IFB-088 in oral capsule divided into 2 doses of 25.0mg administered with 250ml of water at room temperature, seperated by an interval of 12h, in the morning around 8:00am, an in the evening around 8:00pm, for 14 days.
  IFB-088 (15.0-50.0mg) oral capsule: MAD phase: multiple doses of IFB-088 (15.0-50.0mg) will be administered daily during 14 days, in two intakes, separated by an interval of 12 hours.
Arm/Group | SAD IFB-088 2.5mg | SAD IFB-088 5.0mg | SAD IFB-088 10.0mg | SAD IFB-088 20.0mg | SAD IFB-088 40.0mg | SAD IFB-088 60.0mg | MAD IFB-088 15.0mg | MAD IFB-088 30.0mg | MAD IFB-088 50.0mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/ml
  Cmax Dose 1 | 0.54 (34.5) | 0.45 (62.3) | 1.19 (75.5) | 1.39 (16.3) | 2.93 (35.2) | 4.26 (46.3) | 1.70 (87.1) | 2.52 (54.0) | 4.38 (49.8)
  Cmax Dose 2: number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  Cmax Dose 2 |  | 0.37 (59.7) | 1.13 (44.2) | 1.52 (34.3) | 2.39 (31.2) | 4.52 (50.6) | 1.61 (47.2) | 3.58 (41.1) | 6.92 (52.3)

4. Secondary Outcome: Pharmacokinetic: Time to Reach the Maximum Concentration in Plasma (Tmax)
Description: as for outcome 3
Time Frame: Starting 1 hour prior to dosing on Day 1 and until 72 hours after last dosing (Day 17)
Population: 6 patients per cohort have received the verum and are presented. In all groups but one, patients received the verum twice daily. Tmax has hence been measured twice. In the SAD IFB-088 2.5mg cohort, 0 patient received dose 2 as only 1 dose (dose 1) of 2.5mg was given to the patient therefore Tmax Dose 2 has not been measured.
Measure: Median (Inter-Quartile Range); unit: h
Arm/Group | SAD IFB-088 2.5mg | SAD IFB-088 5.0mg | SAD IFB-088 10.0mg | SAD IFB-088 20.0mg | SAD IFB-088 40.0mg | SAD IFB-088 60.0mg | MAD IFB-088 15 mg | MAD IFB-088 30 mg | MAD IFB-088 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
h
  Tmax Dose 1 | 1.5 [1.0 to 1.5] | 1.5 [0.7 to 2.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0] | 1.0 [0.7 to 2.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Tmax Dose 2: number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  Tmax Dose 2 |  | 2.0 [1.0 to 4.0] | 2.0 [2.0 to 2.0] | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 2.0 [0.5 to 4.0] | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0] | 2.0 [1.0 to 3.0]

5. Secondary Outcome: Pharmacokinetic: Terminal Half-life (t1/2)
Description: as for outcome 3
Time Frame: Starting 1 hour prior to dosing on Day 1 and until 72 hours after last dosing (Day 17)
Measure: Mean (Standard Deviation); unit: h
Arm/Group | SAD IFB-088 2.5mg | SAD IFB-088 5.0mg | SAD IFB-088 10.0mg | SAD IFB-088 20.0mg | SAD IFB-088 40.0mg | SAD IFB-088 60.0mg | MAD IFB-088 15 mg | MAD IFB-088 30 mg | MAD IFB-088 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
h | 4.64 (33.3) | 4.61 (56.5) | 5.92 (33.8) | 6.21 (26.9) | 5.76 (10.8) | 5.17 (11.8) | 6.97 (33.1) | 5.70 (22.9) | 6.34 (28.7)

6. Secondary Outcome: Pharmacokinetic: Area Under Plasma Concentration-time Curve From Hour 0 to Last Sample With Measurable Plasma Concentrations (AUClast)
Description: as for outcome 3
Time Frame: Starting 1 hour prior to dosing on Day 1 and until 72 hours after last dosing (Day 17)
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | SAD IFB-088 2.5mg | SAD IFB-088 5.0mg | SAD IFB-088 10.0mg | SAD IFB-088 20.0mg | SAD IFB-088 40.0mg | SAD IFB-088 60.0mg | MAD IFB-088 15 mg | MAD IFB-088 30 mg | MAD IFB-088 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng*h/mL | 2.25 (50.6) | 3.80 (95.2) | 12.5 (47.9) | 17.4 (41.7) | 27.4 (32.5) | 51.1 (40.0) | 18.7 (49.5) | 40.8 (35.7) | 77.2 (48.8)

7. Secondary Outcome: Pharmacokinetic: Apparent Volume of Distribution (Vd/F)
Description: as for outcome 3
Time Frame: Starting 1 hour prior to dosing on Day 1 and until 72 hours after last dosing (Day 17)
Population: 6 patients per cohort have received the verum and are presented. In all groups but one (SAD IFB-088 2.5mg), patients received the verum twice daily. Data were not collected for the SAD IFB-088 2.5 and 5.0mg cohorts
Measure: Mean (Standard Deviation); unit: L
Arm/Group | SAD IFB-088 2.5mg | SAD IFB-088 5.0mg | SAD IFB-088 10.0mg | SAD IFB-088 20.0mg | SAD IFB-088 40.0mg | SAD IFB-088 60.0mg | MAD IFB-088 15 mg | MAD IFB-088 30 mg | MAD IFB-088 50 mg
Number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 6 | 6 | 6 | 6
L |  |  | 5093 (16.9) | 10055 (33.2) | 10408 (16.4) | 10550 (65.5) | 8916 (41.1) | 6860 (43.0) | 7042 (54.5)

8. Secondary Outcome: Pharmacokinetic: Apparent Total Body Clearance (CL/F)
Description: Plasma samples are collected:
  SAD phase - cohort 1 (one intake for daily administration): Day 1 at predose, 0.16, 0.33, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 24, 32h
  SAD phase - cohort 2 to 6 (two intakes for daily administration): Day 1 at predose, 0.33, 0.66, 1, 2, 3, 4, 5, 12, 12.25, 12.5, 13, 14, 16, 18, 24, 32h
  MAD phase (two intakes for daily administration): Day 1 and Day 14 at predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 13, 14, 17, 19 and 21h ; Day 2 (24 hours); Day 7 (predose, 1h and 2 h post dose); Day 15 (24, 30, 36 and 42 hours after Day 14); Day 16 (48, 60 hours after Day 14).
Time Frame: Starting 1 hour prior to dosing on Day 1 and until 72 hours after last dosing (Day 17)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | SAD IFB-088 2.5mg | SAD IFB-088 5.0mg | SAD IFB-088 10.0mg | SAD IFB-088 20.0mg | SAD IFB-088 40.0mg | SAD IFB-088 60.0mg | MAD IFB-088 15 mg | MAD IFB-088 30 mg | MAD IFB-088 50 mg
Number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 6 | 6 | 6 | 6
L/h |  |  | 736 (43.0) | 1146 (45.1) | 1279 (13.9) | 1388 (61.6) | 926 (34.7) | 826 (38.3) | 843 (28.0)

9. Secondary Outcome: Pharmacokinetic: Renal Clearance (CLr)
Description: Urine samples are collected:
  SAD phase - cohort 1 (one intake for daily administration): Day 1 at predose, 0-4 hours, 4-8 hours, 8-16 hours,16-32 hours SAD phase - cohort 2 to 6 (two intakes for daily administration): Day 1 at predose, 0-4, 4-8, 8-12, 12-24, 24-32 hours MAD phase (two intakes for daily administration): Day 1 and Day 14: predose, 0-4, 4-12, 12-24 hours; Day 6: predose, 0-4 and 4-12 hours; Day 15: 24-36, 36-48 hours after Day 14
Time Frame: Starting 1 hour prior to dosing on Day 1 and until 48 hours after last dosing (Day 16)
Population: Data were not collected for the SAD IFB-088 2.5 mg cohort
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | SAD IFB-088 2.5mg | SAD IFB-088 5.0mg | SAD IFB-088 10.0mg | SAD IFB-088 20.0mg | SAD IFB-088 40.0mg | SAD IFB-088 60.0mg | MAD IFB-088 15 mg | MAD IFB-088 30 mg | MAD IFB-088 50 mg
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
mL/min |  | 167 (55.8) | 75.3 (44.6) | 117 (22.3) | 106 (32.4) | 60.5 (37.6) | 76.6 (34.0) | 84.4 (45.0) | 66.2 (36.4)

10. Secondary Outcome: Pharmacokinetic: Percent of Drug Recovered in Urine (Ae %Dose)
Description: as for outcome 9
Time Frame: Starting 1 hour prior to dosing on Day 1 and until 48 hours after last dosing (Day 16)
Population: 6 patients per cohort have received the verum and are presented. In all groups but one (SAD IFB-088 2.5mg), patients received the verum twice daily. Data were not collected for the SAD IFB-088 2.5 cohort
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | SAD IFB-088 2.5mg | SAD IFB-088 5.0mg | SAD IFB-088 10.0mg | SAD IFB-088 20.0mg | SAD IFB-088 40.0mg | SAD IFB-088 60.0mg | MAD IFB-088 15 mg | MAD IFB-088 30 mg | MAD IFB-088 50 mg
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
mg/day |  | 0.52 (67.7) | 0.55 (49.6) | 0.61 (46.2) | 0.44 (44.9) | 0.29 (39.7) | 0.61 (52.5) | 0.74 (56.8) | 0.63 (39.7)

11. Secondary Outcome: Number of Participants With Clinically Significant Change in Physical Evaluation During the Study
Description: the following parameters are assessed during the physical evaluation visit: Cardiovascular system (see specific outcome measure), Digestive system (included spleen organ), alcohol consumption (Ethylotest), General condition, Liver and biliary tracts, Lymphatic system, Muco-cutaneous system, Neck/Thyroide, Nervous system, ENTsystem, Respiratory system, Visual system
Time Frame: SAD & MAD phases: Screening; Day 2 (SAD) or Day 17 (MAD); and at End of study visit (7 to 14 days after last dosing)
Measure: Count of Participants; unit: Participants
Arm/Group | SAD IFB-088 2.5mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Participants
  cardiavascular system | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  digestive system | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  general condition | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  liver and biliary tract | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  lymphatic system | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  muco-cutaneous system | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ENT system | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  respiratory system | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  visual system | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants with no clinically significant changes | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 5 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2

12. Secondary Outcome: Number of Participants With Clinically Significant Change in Physiological Parameters During the Study
Description: Weight measured in kg and height measured in cm, were taken and Body Mass Index was calculated using those 2 values
Time Frame: SAD & MAD phases: Screening; Day 2 (SAD) or Day 17 (MAD); and at End of study visit (7 to 14 days after last dosing)
Measure: Count of Participants; unit: Participants
Arm/Group | SAD IFB-088 2.5mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Participants
  Number of subjects with clinically significant change in weight | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of participants with clinically significant change in BMI | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants without clinically significant changes | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2

13. Secondary Outcome: Number of Participants With With Clinically Significant Change in Cardiovascular Functions During the Study
Description: This safety outcome aims at monitoring cardiovascular functions and identify potential adverse events/reactions (clinical assessment combined with ECGs and vital signs assessments).
Time Frame: From screening visit until end of study visit (7 to 14 days after last dosing)
Measure: Count of Participants; unit: Participants
Arm/Group | SAD IFB-088 2.5mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Participants
  Number of participants with clinically significant change in electrocardiogram parameters (ECG) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of participants with no clinically significant changes in ECG | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2

14. Secondary Outcome: Number of Participants With With Clinically Significant Change in Tympanic Body Temperature During the Study
Description: Tympanic body temperature will be measured at the time frame described underneath.at the following Timepoints :
  change in body temperature (fever) will be reported per patient per group.
Time Frame: SAD phase (cohorts 1 to 6):Screening, Day -1;Day 1 ;end (7 to 14 days after last dosing) MAD phase: Screening;Day -1; Day 1 ;predose at Day 2, Day 4, Day 6, Day 8, Day 10, Day 12; Day 14 ; Day 17; end (7 to 14 days after last dosing)
Measure: Count of Participants; unit: Participants
Arm/Group | SAD IFB-088 2.5mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Participants
  Nr of participants presenting clinically significant change in tympanic body temp. during the study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nr of participants without clinically significant change in tympanic body temp. throughout the study | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2

15. Secondary Outcome: Number of Participants With With Clinically Significant Change in Hematology Parameters During the Study
Description: This safety outcome aims at monitoring hematology parameters:
  Red blood cell (RBC) count, hemoglobin, hematocrit, white blood cell (WBC) count (neutrophils, lymphocytes, monocytes, eosinophils, basophils), platelets, reticulocyte count will be monitored from screening to end of study visit (7 to 14 days after last dosing), at several time points.
  When a participant experienced clinically significant change in the parameter, at least once during the study, he/she is recorded in the table.
Time Frame: SAD phase: Screening; Day -1; Day 2 (24 hours); end of study visit (7 to 14 days after last dosing) MAD phase: Screening; Day -1; predose, at Day 3, Day 6, Day 10, Day 13; Day 17; end of study visit (7 to 14 days after last dosing)
Measure: Count of Participants; unit: Participants
Arm/Group | SAD IFB-088 2.5mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Participants
  Number of participants with clinically significant changes in eosinophils at one timepoint | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of participants with clinically significant changes in haemoglobin at one timepoint | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of participants with clinically significant changes in haematocrit at one timepoint | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of participants with clinically significant changes in lymphocytes at one timepoint | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of participants with clinically significant changes in monocytes at one timepoint | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of participants with clinically significant changes in neutrophils at one timepoint | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of participants with clinically significant changes in platelets at one timepoint | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of participants with clinically significant changes in reb blood cells at one timepoint | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of participants with clinically significant changes in reticulocytes at one timepoint | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of participants with clinically significant changes in leucocytes at one timepoint | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of participants with clinically significant changes in white blood cells at one timepoint | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nr of participants without clinically significant changes in hematology param. throughout the study | 6 | 2 | 6 | 2 | 4 | 2 | 6 | 2 | 5 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2

16. Secondary Outcome: Number of Participants With With Clinically Significant Change in Coagulation Parameters During the Study
Description: This safety outcome aims at monitoring coagulation parameters such as Activated partial thromboplastin time (APTT), international normalized ratio (INR)
Time Frame: SAD phase: Screening; Day -1; Day 2 (24 hours); end of study visit (7 to 14 days after last dosing) MAD phase: Screening; Day -1; predose at Day 3, Day 6, Day 10, Day ; Day 17; end of study visit (7 to 14 days after last dosing)
Measure: Count of Participants; unit: Participants
Arm/Group | SAD IFB-088 2.5mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Participants
  number of participants with clinically significant changes in INR during the study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants with clinically significant changes in APTT during the study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants without clinically significant changes in coagulation throughout the study | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2

17. Secondary Outcome: Number of Participants With With Clinically Significant Change in Blood Biochemistry Parameters During the Study
Description: This safety outcome aims at monitoring the following blood biochemistry parameters:
  Sodium, potassium, chloride, calcium, total bilirubin, alanine aminotransferase (ASAT), aspartate aminotransferase (ALAT), gamma-glutamyl transferase (GGT), alkaline phosphatases, total protein, albumin, urea, uric acid, bicarbonate, creatine phosphokinase (CPK), creatinine, glycaemia, lactate dehydrogenase (LDH), total cholesterol, HDL and LDL cholesterol, triglycerides
Time Frame: SAD phase: Screening; Day -1; Day 2 (24 hours); end of study visit (7 to 14 days after last dosing) MAD phase: Screening; Day -1; predose at Day 3, Day 6, Day 10, Day 13; Day 17; end of study visit (7 to 14 days after last dosing)
Measure: Count of Participants; unit: Participants
Arm/Group | SAD IFB-088 2.5mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Participants
  number of participants with clinically significant changes in ion (Na, K, Cl, Ca, HCO3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants with clinically significant changes in aminotransferases (ASAT, ALAT, GGT) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants with clinically significant changes in cholesterol (total, HDL, LDL) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants with clinically significant changes in triglycerides | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants with clinically significant changes in glycaemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants with clinically significant changes in total bilirubin | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants with clinically significant changes in alkaline phosphatases | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants with clinically significant changes in total protein | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants with clinically significant changes in albumin | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants with clinically significant changes in urea and uric acid | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nr of participants with clinically significant changes in creatinine and creatinine phosphokinase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants with clinically significant changes in lactate dehydrogenase (LDH) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nr of participants without clinically significant changes in biochem. param. throughout the study | 6 | 2 | 5 | 1 | 5 | 2 | 6 | 1 | 6 | 2 | 4 | 2 | 6 | 2 | 6 | 2 | 6 | 2

18. Secondary Outcome: Number of Participants With Clinically Significant Change in Urinary Functions/Parameters During the Study
Description: This safety outcome aims at monitoring urinary functions/parameters:
  Specific gravity, pH, glucose, protein, blood, nitrites, leucocytes and ketones by dipstick.
  Results are given as "absent" or "present, not clinically significant" or "present clinically significant".
  A cytobacteriological exam will be done if abnormal results on dipstick). Beta 2 microglobulin (B2M), proteinuria and creatinuria will be also monitored.
Time Frame: SAD phase: Screening; Day -1; Day 1 (predose, 12, 24, 32 hours); end of study visit (7 to 14 days after last dosing) MAD phase: Screening; Day -1; predose at Day 1, Day 3, Day 6, Day 10, Day 13; Day 17; end of study visit (7 to 14 days after last dosing)
Measure: Count of Participants; unit: Participants
Arm/Group | SAD IFB-088 2.5mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Participants
  Nr of participants with clinically significant change of parameters present on dispstick (see above) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants with clinically significant changes of beta2 microglobulin | 0 | 0 | 0 | 0 | 00 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants with clinically significant changes of proteinuria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants with clinically significant changes of creatinuria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants without clinically significant changes of urinary parameters | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2

19. Secondary Outcome: Number of Participants With Clinically Significant Change in Vigilance and Mood During the Study
Description: Assessment and monitoring of the vigilance/mood of healthy volunteers through the use of a Bond-Lader Visual Analogue Scale listing 16 mood items, with 2 words at the beginning and the end of the scale bar. Depending on the item, the scale would go from better to worse (ie strong to weak) or the opposite (Hostile to friendly). Alertness, Self-contentment, Calmness are computed by averaging their respective items and are mentionned in the volunteer file.
Time Frame: SAD Phase: Screening; Day 1 (predose, 1.5, 12, 32 hours) MAD Phase: Screening; Day 1 (predose, 1.5, 12 hours); Day 14 (predose, 1.5, 12 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | SAD IFB-088 2.5mg | SAD Placebo 2.5mg | SAD IFB-088 5.0mg | SAD Placebo 5.0mg | SAD IFB-088 10.0mg | SAD Placebo 10.0mg | SAD IFB-088 20.0mg | SAD Placebo 20.0mg | SAD IFB-088 40.0mg | SAD Placebo 40.0mg | SAD IFB-088 60.0mg | SAD Placebo 60.0mg | MAD IFB-088 15.0mg | MAD Placebo 15.0mg | MAD IFB-088 30.0mg | MAD Placebo 30.0mg | MAD IFB-088 50.0mg | MAD Placebo 50.0mg
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Participants
  number of participants with clinically significant changes of vigilance or mood during the study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  number of participants without clinically significant changes of vigilance or mood during the study | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2

20. Other Pre Specified Outcome: SAD Exploratory Biomarkers Analysis
Description: Blood samples will be collected and stored in a biobank to explore potential biomarkers that remain to be identified
Time Frame: SAD phase: Day 1 at predose, 1.5 hours and 24 hours
Reporting Status: Not Posted

21. Other Pre Specified Outcome: MAD Exploratory Biomarkers Analysis
Description: Blood samples will be collected and stored in a biobank to explore potential biomarkers that remain to be identified
Time Frame: MAD phase: Day 1 and Day 14 at predose, 1.5 hours and 24 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 18 months
Description: Safety was the primary endpoint of this Phase 1 study Number of participants with TEAE are reported in the primary endpoint section. As this section is more appropriate to describe TEAE, it was decided to further describe the primary endpoint in this section.
Groups:
- SAD IFB-088 2.5mg: cohort 1: single daily dose of 2.5mg IFB-088 oral capsule, administered in the morning (8:00am), in one intake
- SAD IFB-088 5.0mg: cohort 2: single daily dose of 5.0mg IFB-088 oral capsule, administered in two intakes of 2.5mg, 12 hours apart, in the morning (8:00am), and in the evening (8:00pm)
- SAD IFB-088 10.0mg: cohort 3: single daily dose of 10.0mg IFB-088 oral capsule, administered in two intakes of 5.0mg, 12 hours apart, in the morning (8:00am), and in the evening (8:00pm)
- SAD IFB-088 20.0mg: cohort 4: single daily dose of 20.0mg IFB-088 oral capsule, administered in two intakes of 10.0mg, 12 hours apart, in the morning (8:00am), and in the evening (8:00pm)
- SAD IFB-088 40.0mg: cohort 5: single daily dose of 40.0mg IFB-088 oral capsule, administered in two intakes of 20.0mg, 12 hours apart, in the morning (8:00am), and in the evening (8:00pm)
- SAD IFB-088 60.0mg: cohort 6: single daily dose of 60.0mg IFB-088 oral capsule, administered in two intakes of 30.0mg, 12 hours apart, in the morning (8:00am), and in the evening (8:00pm)
- SAD Placebo: (cohort 1 to 6): single daily dose of placebo oral capsule, administered in two intakes (except for the first SAD dose that is administered in one intake), at 12h intervals, in the morning (8:00am) and in the evening (8:00pm)
- MAD IFB-088 15.0mg: cohort 7: subject taking 15.0mg of IFB-088 oral capsule divided in two dose of 7.5mg, at an interval of 12h, in the morning (8:00am), and in the evening (8:00pm), for 14 days.
- MAD IFB-088 30.0mg: cohort 8: subject taking 30.0mg of IFB-088 oral capsule divided in two dose of 15.0mg, at an interval of 12h, in the morning (8:00am), and in the evening (8:00pm), for 14 days.
- MAD IFB-088 50.0mg: cohort 9: subject taking 50.0mg of IFB-088 oral capsule divided in two dose of 25.0mg, at an interval of 12h, in the morning (8:00am), and in the evening (8:00pm), for 14 days.
- MAD Placebo: (cohort 7 to 9): subject taking placebo oral capsule divided in two doses, at an interval of 12h, in the morning (8:00am), and in the evning (8:00pm), for 14 days.
Arm/Group | SAD IFB-088 2.5mg | SAD IFB-088 5.0mg | SAD IFB-088 10.0mg | SAD IFB-088 20.0mg | SAD IFB-088 40.0mg | SAD IFB-088 60.0mg | SAD Placebo | MAD IFB-088 15.0mg | MAD IFB-088 30.0mg | MAD IFB-088 50.0mg | MAD Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 2/6 | 2/6 | 2/6 | 3/6 | 2/12 | 4/6 | 1/6 | 4/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAD IFB-088 2.5mg (N=6) | SAD IFB-088 5.0mg (N=6) | SAD IFB-088 10.0mg (N=6) | SAD IFB-088 20.0mg (N=6) | SAD IFB-088 40.0mg (N=6) | SAD IFB-088 60.0mg (N=6) | SAD Placebo (N=12) | MAD IFB-088 15.0mg (N=6) | MAD IFB-088 30.0mg (N=6) | MAD IFB-088 50.0mg (N=6) | MAD Placebo (N=6)
headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
catheter site related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
pollakyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT03610334/Prot_SAP_000.pdf